CLINICAL TRIAL: NCT03509415
Title: Reflectance Confocal Microscopy to Diagnose Basal Cell Carcinoma
Brief Title: Reflectance Confocal Microscopy to Diagnose BCC
Status: Completed | Type: Observational
Sponsor: Skin Care Network Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HS-MAV-003
Record Dates: First submitted 2018-04-16; First posted 2018-04-26 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Basal Cell Carcinoma
Keywords: Confocal; RCM; Imaging; Skin cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms | interventions — Intravital Microscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: In-vivo imaging — Skin cancer is imaged using RCM and a diagnosis is recorded before patient is returned to standard of care (biopsy).

SUMMARY:
It is proposed to undertake a study to determine the diagnostic utility of using RCM for the diagnosis of Basal Cell Carcinoma (BCC) in a tertiary referral centre as outlined by the recent NICE report (Nov 2015). This will allow an assessment of the potential to avoid diagnostic biopsy within the treatment pathway.

DETAILED DESCRIPTION:
Study Design This is an observational, non-randomised, non-controlled, prospective cohort study to look at the efficacy of in vivo RCM as a diagnostic tool in the diagnosis of BCC.

Study Hypothesis The hypothesis of this study is that the use of RCM is would enable a reduction in the number of diagnostic biopsies taken before definitive treatment of BCC by at least 50%.

The secondary hypothesis is that the intra- & inter-observer agreement for interpreting the RCM images will have kappa scores 0.6 or greater (indicating good agreement).

Patients will be recruited from the outpatient clinic of Skin Care Network London.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Patient suspected of having a primary basal cell carcinoma that is a candidate for surgical treatment.
3. Patient willing and able to give informed consent

Exclusion Criteria:

1. Recurrent or other higher-risk BCC
2. Patient with basal cell naevus syndrome
3. Patient treated with hedgehog inhibitor medication (vismodegib)
4. Patient not suitable for diagnostic biopsy
5. Location of lesion unsuitable, inaccessible or impractical for scanning with RCM as determined by investigator
6. Patient with co-morbidities such as other skin disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting at a skin cancer clinic with a lesion that is clinically suspicious for BCC
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | During exam (biopsy results typically available within one week).
  Specificity & Sensitivity of RCM in diagnosing Basal Cell Carcinoma in non-pigmented lesions compared to standard histology

SECONDARY OUTCOMES:
intra- & inter-observer agreement for interpreting the RCM images | 6 months
  A measure of how consistently readers can diagnose from confocal images.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Stevens, MA PhD, Principal Investigator — Skin Care Network Ltd.
Locations (1):
- Skin Care Network Barnet Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stevens HP, Pampena R, Farnetani F, Pellacani G, Angus C, El-Jabbour JN. Reflectance confocal microscopy in diagnosing basal cell carcinoma in the UK: a prospective observational single-centre trial. Br J Dermatol. 2025 Jan 24;192(2):206-214. doi: 10.1093/bjd/ljae356. PMID 39259284

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT03509415/Prot_SAP_000.pdf